CLINICAL TRIAL: NCT05276102
Title: The Effects of Repeated Exposure to Antiseptics During COVID-19 Pandemic on Skin Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Dario Leskur, Assistant professor, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2181-198-03-04-22-0009
Record Dates: First submitted 2022-03-10; First posted 2022-03-11 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Irritation/Irritant; ICD - Irritant Contact Dermatitis; Antiseptic
MeSH Terms: conditions — Dermatitis, Irritant

STUDY DESIGN:
Intervention Model Description: Each volar forearm of the participants will be divided in three sites, with each site randomly assigned to repeated exposure to antiseptic, repeated exposure to deionized water (sham irritation) or will be left intact.
  One forearm will be treated with the commercially available emollient three times a day while the other will be left untreated. Treated forearm (left or right) will be chosen according to randomization protocol (double randomization).
Who Masked: Investigator, Outcomes Assessor
Masking Description: One forearm will be treated with the commercially available emollient while the other will be left untreated. Therefore the participants will not be blinded but the outcomes assessor and the principal investigator will be blinded to the treatment.
  Disinterested third party will perform the randomization and treatment allocation, as well as keep the code breaks in case of medical emergency or adverse events of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Repated exposure to antiseptic and treatment (Active Comparator): Repeated exposure of forearm skin to antiseptic (once daily for 2 hours under occlusion, during three weeks) Emollient cream treatment 3 times a day
  Interventions: Other: Emollient cream
- Sham irritation and treatment (Active Comparator): Repeated exposure of forearm skin to deionized water (once daily for 2 hours under occlusion, during three weeks) Emollient cream treatment 3 times a day
  Interventions: Other: Emollient cream
- No irritation and treatment (Active Comparator): Intact skin on forearms Emollient cream treatment 3 times a day
  Interventions: Other: Emollient cream
- Repated exposure to antiseptic and no treatment (No Intervention): Repeated exposure of forearm skin to antiseptic (once daily for 2 hours under occlusion, during three weeks) No emollient cream treatment
- Sham irritation and no treatment (No Intervention): Repeated exposure of forearm skin to deionized water (once daily for 2 hours under occlusion, during three weeks) No emollient cream treatment
- No irritation and no treatment (No Intervention): Intact skin on forearms No emollient cream treatment

INTERVENTIONS:
Other: Emollient cream — Commercially available emollient cream
  Arms: No irritation and treatment; Repated exposure to antiseptic and treatment; Sham irritation and treatment

SUMMARY:
The global coronavirus disease pandemic (COVID-19) has led to an increased need to wear protective equipment such as wearing face masks and practicing hygiene measures such as more frequent use of antiseptics. These measures can lead to changes in the skin, the development of new inflammatory skin diseases or exacerbation of existing ones, with health professionals especially under the risk of developing these changes. Changes in the skin of the hands due to the use of antiseptics have been observed in a number of studies, however, part of the study was based solely on subjects' self-assessment or clinical assessment of researchers, and only a small part on objective measurements of skin parameters. Also, the impact of prolonged use of antiseptics and the impact of measures to prevent and protect against irritation such as topical application of emollient preparations have not been investigated.

The impact of repeated use of antiseptics in the repeated exposure model on the forearms will be investigated. This model is a modification of the existing model of irritative dermatitis induced by sodium lauryl sulfate where the original irritant was replaced by an antiseptic solution.

ELIGIBILITY:
Inclusion Criteria:

* young, healthy volunteers who gave written informed consent

Exclusion Criteria:

* skin disease, skin damage on measurement sites
* use of corticosteroids, antihistamines and immunomodulators a month prior the inclusion and during the trial
* use of emollients three days prior the inclusion in the trial
* non-adherence to the trial protocol
* pregnancy and lactation
* skin cancer
* immunosuppression
* exposure to artificial UV radiation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Transepidermal water loss change | Baseline value measurements on the first day of trial, during the three weeks the skin is repeatedly exposed to antiseptic as well recovery during the following two weeks
  Tewameter will be used to assess skin barrier function as a measurement of the water loss (g/hm2).
Stratum corneum hydration change | Baseline value measurements on the first day of trial, during the three weeks the skin is repeatedly exposed to antiseptic as well recovery during the following two weeks
  Corneometer will be used to estimate skin dryness. It is a relative measurement and uses arbitrary units (AU).
Erythema change | Baseline value measurements on the first day of trial, during the three weeks the skin is repeatedly exposed to antiseptic as well recovery during the following two weeks
  Mexameter will be used to assess erythema. It is a relative measurement and uses arbitrary units (AU).
Melanin content change | Baseline value measurements on the first day of trial, during the three weeks the skin is repeatedly exposed to antiseptic as well recovery during the following two weeks
  Mexameter will be used to assess skin melanin content. It is a relative measurement and uses arbitrary units (AU).
Clinical score | Baseline value measurements on the first day of trial, during the three weeks the skin is repeatedly exposed to antiseptic as well recovery during the following two weeks
  Skin response to irritation and treatment will be assessed using a five-point scale (0, 1/2, 1, 2 and 3) to describe changes in skin erythema, roughness, scaling, oedema, and fissures, with higher score signifying a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Montero-Vilchez T, Cuenca-Barrales C, Martinez-Lopez A, Molina-Leyva A, Arias-Santiago S. Skin adverse events related to personal protective equipment: a systematic review and meta-analysis. J Eur Acad Dermatol Venereol. 2021 Oct;35(10):1994-2006. doi: 10.1111/jdv.17436. Epub 2021 Jun 29. PMID 34077565
- [Background] Akl J, El-Kehdy J, Salloum A, Benedetto A, Karam P. Skin disorders associated with the COVID-19 pandemic: A review. J Cosmet Dermatol. 2021 Oct;20(10):3105-3115. doi: 10.1111/jocd.14266. Epub 2021 Jul 1. PMID 34077629
- [Background] Elston DM. Occupational skin disease among health care workers during the coronavirus (COVID-19) epidemic. J Am Acad Dermatol. 2020 May;82(5):1085-1086. doi: 10.1016/j.jaad.2020.03.012. Epub 2020 Mar 18. No abstract available. PMID 32171807
- [Background] Park SR, Han J, Yeon YM, Kang NY, Kim E. Effect of face mask on skin characteristics changes during the COVID-19 pandemic. Skin Res Technol. 2021 Jul;27(4):554-559. doi: 10.1111/srt.12983. Epub 2020 Nov 20. PMID 33217053
- [Background] Tupker RA, Willis C, Berardesca E, Lee CH, Fartasch M, Agner T, Serup J. Guidelines on sodium lauryl sulfate (SLS) exposure tests. A report from the Standardization Group of the European Society of Contact Dermatitis. Contact Dermatitis. 1997 Aug;37(2):53-69. doi: 10.1111/j.1600-0536.1997.tb00041.x. PMID 9285167